CLINICAL TRIAL: NCT07136350
Title: The Relationship of Nurse Caring Communication Engagement and Patient's Satisfaction With Readmission Rates
Brief Title: Nurse Caring Communication Engagement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Florida Atlantic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2352402
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-07

CONDITIONS: Perceptions of Caring; Hospital Readmissions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication Coaching + S.M.A.R.T. Discharge Tool (Experimental): Nurses in this group will receive caring communication coaching (2 CEUs) and implement the S.M.A.R.T. discharge tool. Outcomes will be assessed at T0, T1 (4 weeks), and T2 (1 month post-T1).
  Interventions: Other: Communication Coaching; Behavioral: Implement S.M.A.R.T. Discharge Tool
- Control Group (No Intervention): Nurses in this group will continue standard discharge practices without coaching or the S.M.A.R.T. tool. Outcomes will be assessed at the same time points (T0, T1, T2).

INTERVENTIONS:
Other: Communication Coaching — Nurses in this group will receive caring communication coaching (2 CEUs).
  Arms: Communication Coaching + S.M.A.R.T. Discharge Tool
Behavioral: Implement S.M.A.R.T. Discharge Tool — Implement the S.M.A.R.T. discharge tool.
  Arms: Communication Coaching + S.M.A.R.T. Discharge Tool

SUMMARY:
The overall goal will be to explore the effectiveness of caring communication coaching with the implementation of a discharge tool in the acute care setting and its impact on the nurse-patient relationship. Integrating communication strategies through a caring lens with an educational tool will seek to address the missing components that satisfy patient care experience, satisfaction with care, prevention of complications, reduction of readmission rates, and improved outcomes. This study will evaluate how these interventions can narrow the gap in the literature and enhance the quality of patient care which can ultimately improve health outcomes.

ELIGIBILITY:
Patient inclusion criteria 1. 18 years or older; inpatient admission to the hospital. 2. Speak, read, write, and understand English. Nurse inclusion criteria

1. Works at Baptist Health South Florida hospital system and provides direct bedside patient care.
2. Have an active Florida Nurses license.
3. Registered Nurse (AA, BSN, MSN).

Exclusion criteria: The exclusion criteria are:

Patient Exclusion criteria

1. Hospice and psych patients.
2. Unable to commit to the interview. Nurse Exclusion criteria

1. Director, managers, charge nurse/relief charge nurse. 2. Nurses floated to the unit 3. Unable to commit to the interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Nurse Caring Behaviors (Patient-Perceived) | 2 months
  Assessed using a validated patient questionnaire, the five-item Watson's Caritas of Human Caring (WCHC) - At discharge (T0), and follow-ups at T1 and T2
Sustained Change in Nurses' Caring Communication Skills (Self-Reported) | 2 months
  Measured using a nurse self-report 18-item survey, the Health Professionals Skills Scale (HP-CSS). Change in nurse scores between T0, T1, and T2 to evaluate long-term impact. - From baseline to 1 month post-intervention (T0 to T2)

SECONDARY OUTCOMES:
30-day Hospital Readmission Rate | 2 months
  Overall monthly readmission rates (frequency) for the departments included in the study - 30-day readmission is defined as a patient who is re-admitted to the hospital within 30 days or less from their last hospital discharge date.

CONTACTS AND LOCATIONS:
Locations (1):
- Baptist Hospital of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No